CLINICAL TRIAL: NCT01290913
Title: Xolair Enhances Oral Desensitization in Peanut Allergic Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lynda Schneider (Other)
Responsible Party: Sponsor-Investigator, Lynda Schneider, Associate Professor, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHB10090470; Xolair and Peanut Allergy (Other Grant/Funding Number: TRF)
Record Dates: First submitted 2011-02-04; First posted 2011-02-07 (Estimated); Results first posted 2015-02-20 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Peanut Allergy
Keywords: peanut allergy; Xolair
MeSH Terms: conditions — Peanut Hypersensitivity | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- omalizumab, oral desensitization (Experimental): Patients receive omalizumab along with oral peanut desensitization.
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Omalizumab — Omalizumab is an antibody that helps decrease allergic responses in the body
  Other Names: Xolair

SUMMARY:
This is a pilot feasibility study, using Xolair pretreatment for oral peanut desensitization.

DETAILED DESCRIPTION:
We hypothesize that pretreatment with anti-IgE mAb will greatly reduce the side effects and allergic reactions that occur during oral desensitization to peanut and will enhance the development of oral tolerance in patients with severe peanut allergy.

We will follow the patients for 5 years following study completion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with severe peanut allergy, between the ages of 7-25 years, having a history of significant clinical symptoms within 1 hr of peanut ingestion.
2. Total IgE >50 kU/L but <2,0000 kU/L.
3. Sensitivity to peanut will be documented by a positive skin prick test result and RAST test to peanut, with 20 kU/L as a lower limit for eligibility.
4. Patients must also fail a double blind food challenge with peanut at a dose of 100 mg or less (after a cumulative dose of 186 mg), with minimal or no reactions to the placebo challenge.
5. All female subjects of childbearing potential will be required to provide a urine sample for pregnancy testing that must be negative one week before being allowed to participate in the study.
6. Subjects must be planning to remain in the study area during the trial.
7. Subjects and/or their parents must be trained on the proper use of the Epi-Pen to be allowed to enroll in the study.

Exclusion Criteria:

Due to the risk of serious systemic anaphylactic reactions to peanut in this study, we will exclude:

1. Patients with acute infections, autoimmune disease, severe cardiac disease, and those who are treated with beta-adrenergic antagonistic drugs (beta-blockers, which increase the risk of more serious symptoms of anaphylaxis).
2. Subjects having a history of severe anaphylaxis to peanut requiring intubation or admission to an ICU, frequent urticaria, or history consistent with poorly controlled persistent asthma.
3. Total IgE > 2,000 IU/mL.
4. Subjects with unstable angina, significant arrhythmia, uncontrolled hypertension, chronic sinusitis, or other chronic or immunological diseases that in the mind of the investigator might interfere with the evaluation or administration of the test drug or pose additional risk to the subject e.g. gastrointestinal or gastroesophageal disease, chronic infections, scleroderma, hepatic and gallbladder disease, chronic non-allergic pulmonary disease.
5. Subject with an FEV1 or PEF less than 80% predicted with or without controller medication (if able to perform the maneuver) at screening, the oral desensitization visit, or food challenge visit.
6. Subjects who have received an experimental drug in the last 30 days prior to admission into this study or who plan to use an experimental drug during the study, who are current users of oral, intramuscular, or intravenous corticosteroids, or tricyclic antidepressants, or who are using medication that could induce adverse gastrointestinal reactions during the study.
7. Subjects refusing to sign the EpiPen Training Form.
8. Pregnant or breast-feeding females.
9. Subjects with severe food associated eczema, dermatitis herpetiformis, eosinophilic esophagitis, eosinophilic enteritis, proctocolitis, food protein induced enterocolitis syndrome (FPIES) or other gastrointestinal diseases. These requirements are necessary to limit the study to patients with primarily IgE mediated peanut allergy, and to exclude patients with peanut sensitivity mediated by cellular/T cell (non-IgE mediated) mechanisms.

Ages: 7 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2011-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rima T Rachid, MD, Principal Investigator — Children's Hospital, Harvard Medical School; Lynda Schneider, MD, Study Director — Children's Hospital, Harvard Medical School
Locations (1):
- Children's Hospital Boston, Harvard Medical School, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Abdel-Gadir A, Schneider L, Casini A, Charbonnier LM, Little SV, Harrington T, Umetsu DT, Rachid R, Chatila TA. Oral immunotherapy with omalizumab reverses the Th2 cell-like programme of regulatory T cells and restores their function. Clin Exp Allergy. 2018 Jul;48(7):825-836. doi: 10.1111/cea.13161. Epub 2018 May 29. PMID 29700872

RESULTS

PARTICIPANT FLOW:
Groups:
- Omalizumab, Oral Desensitization: Omalizumab treatment and oral peanut desensitization
Period: Overall Study
Arm/Group | Omalizumab, Oral Desensitization
Started | 13
Completed | 12
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Omalizumab, Oral Desensitization
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Tolerated Rapid Oral Peanut Desensitization to a Dose of 500 mg Peanut Flour (Cumulative Dose, 1,000 mg)
Description: To tolerate refers to the ability of the patient to ingest the challenge dose of 500 mg peanut flour (1000 mg cumulatively) with either no or mild symptoms.
Time Frame: First day of desensitization
Measure: Number; unit: participants
Arm/Group | Omalizumab, Oral Desensitization
Number analyzed (Participants) | 13
participants | 13

2. Secondary Outcome: Number of Participants That Tolerated Rapid Oral Peanut Desensitization to a Dose of 4,000 mg of Peanut Flour.
Description: To tolerate refers to the ability of the patient to ingest the final challenge of 4000mg peanut flour, with either no or mild symptoms.
Time Frame: after 7-8 wks of desensitization
Measure: Number; unit: participants
Arm/Group | Omalizumab, Oral Desensitization
Number analyzed (Participants) | 13
participants | 12

ADVERSE EVENTS:
Arm/Group | Omalizumab, Oral Desensitization
Serious Adverse Events (participants affected / at risk) | 2/13
Other Adverse Events (participants affected / at risk) | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omalizumab, Oral Desensitization (N=13)
Anaphylaxis (General disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab, Oral Desensitization (N=13)
Allergic Reaction (Immune system disorders) | 10 — Allergic reaction to peanut. 6 of the 13 subjects (46%) had no or a single grade 1 allergic reaction. Six of the 13 patients (39%) experienced a grade 2 or 3 adverse event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No